CLINICAL TRIAL: NCT07281040
Title: Preparatory Work for a Multi-arm, Multi-stage Trial of Adjunctive Treatments in Patients Hospitalised With Heart Failure (Pre-MAMMOTH-HF)
Brief Title: Preparatory Work for a Trial of Adjuncts to Diuretic Treatment in Patients Hospitalised With Heart Failure: Addressing Uncertainties and Building Consensus
Acronym: Pre-MAMMOTH-HF
Status: Recruiting | Type: Observational
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Hull York Medical School (Unknown); University of Birmingham (Other); Robertson Centre for Biostatistics University of Glasgow Glasgow G12 8QQ (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIHR207987
Record Dates: First submitted 2025-09-12; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient and carer panel using nominal group approach and thematic analysis — Patient and carer panel using nominal group approach and thematic analysis

SUMMARY:
Aims and Objectives

1. Choose which adjunctive therapies, at what dose, and for how long
2. Choose the dose(s) of IV furosemide to be used as the comparator
3. Choose primary and secondary outcomes
4. Estimate recruitment and engage sites for a future trial

Work package 2a methods overview

1. An online survey of clinicians (doctors, nurses and pharmacists) assessing potential ability to recruit and the acceptability of each adjunct and willingness to support a trial.
2. Evidence generated (survey and reviews) will be considered by an expert panel (N=20-25) including expert clinicians and allied health professionals who care for people with HF using a modified Delphi approach. The panel will make recommendations on all aspects of the trial design.
3. A patient and carer panel of people with a recent hospitalisation (<6 months) for HF will provide recommendations on trial endpoints. The patient-and-carer advisory group (PCAG) will also input into these discussions.

DETAILED DESCRIPTION:
Online Survey An online survey of clinicians (doctors, nurses and pharmacists) assessing potential ability to recruit and the acceptability of each adjunct and willingness to support a trial. The survey will also engage the clinical community and gain wider input into the acceptability of each adjunctive therapy to inform trial decision making (aims 1,2, 4).

Through the British Society for Heart Failure and its Research Network, the Royal College of Physicians, and through professional networks we will identify sites interested in participating in the survey and engaging with this research project.

We will present the trial's concept and rationale. Interested sites will then be asked to complete an online survey designed using the findings of the above reviews and hosted on the Qualtrics secure online survey platform.

We will seek input from potential trial sites (n~30) about the acceptability of each intervention (for different doses/durations), with the opportunity to provide reasons for acceptability (or lack thereof). Closed questions will assess willingness to randomise and open questions to understand reasons for or against randomisation. The survey will assess interest in participation and give a realistic estimate of the ability of a trial to recruit patients, and hence estimate the time required for any trial. Results will be analysed using descriptive statistics and qualitative content analysis.56

Ethical approval will be obtained from the University of Hull Research Ethics Committee. The questionnaire will be piloted amongst 5-10 healthcare workers who care for patients with HF and oral or written feedback provided. Once amendments have been agreed by the research team the survey will be circulated via the BSH, British Cardiovascular Society, Royal College of Physicians, and professional networks.

The results of the survey will be shared with the expert panel and patient and carer group to inform discussions and decision making. The results will also be submitted as a poster and/or oral abstract to national and international HF and cardiology conferences. Opportunities for written peer reviewed publication will be explored.

Output: Key stakeholders will be informed about the study; we will gain broader insight into the acceptability of different treatments; we will understand the sites likely to be able to host the trial; and we will be able to estimate the potential numbers of patients for trial recruitment to inform our modelling in work package 2b).

Expert panel consensus meetings Evidence generated (systematic and umbrella reviews [WP1], and the online survey) will be considered by an expert panel (N = 20 - 25) including expert clinicians and allied health professionals who care for people with HF using a modified Delphi approach.57 The panel will make recommendations on the uncertainties 1-4 detailed above.

Panellists will include: clinical specialists who have frequent contact with people with HF (HF cardiologists, palliative care, geriatricians, renal physicians, general practitioners), HF nurses, pharmacists, and non-medical prescribers) from across the UK, identified through national societies and charities, and the professional networks of the research team. The primary criterion for being invited to join the group will be expertise in some aspect of HF (e.g. via published work, personal involvement in previous heart failure trials or recommendations from experts in the field).

The group will be chaired by Professor Theresa McDonagh, leader of the International Consortium for Health Outcomes Measurement (ICHOM). A panel of 20-25 members will ensure we maintain representation across specialties and stability of responses over the three rounds of the Delphi.58

A report of the findings from WP1 and online survey will be sent to the expert panel by email at least two weeks before the first meeting. An initial briefing meeting arranged before the first round of voting takes place. Three rounds of decision making are planned (month 8, 9, and 10).

Round 1 - Month 8 The initial meetings will focus on agreeing the adjunctive treatments to take forward. An email delphi survey will use a bespoke rating form to collect initial ratings (out of 10) on the adjuvant treatments under consideration (drug, dose, duration). Email feedback will be provided of own score and group score before the first online meeting. For a treatment option to go forward without discussion, two-thirds of experts must rate it at least 7/10 and none must rate it lower than 5/10. Two-thirds of respondents must rate a treatment option as 4/10 or lower, for it to be dropped without discussion. All other options are for discussion in the online meetings.

Round 2 - Month 9 Two online meetings will be held via MS Teams or Zoom to consider interventions and usual (standard) care. There will be discussion about the interventions where consensus was not reached in the email Delphi in round 1, and decisions regarding interventions will be formally ratified. A definition of usual care to be used in the trial will also be discussed and ratified. Following each online meeting, detailed notes will be circulated confirming decisions made and listing those left to be considered. A second round of voting will take place after the two online meetings, having discussed the evidence and considering other panellists' views.59 Agreement on the recommendations of the interventions (dose, duration, monitoring) and usual care will be reached.

Round 3 A third online meeting will consider outcomes to be used in the trial. Prior to the online meeting, panellists will be sent an email survey containing a list of potential outcomes for the trial, including the existing core outcome set for people with heart failure. Panellists will be asked to rank these using the bespoke rating system described above. The results will be discussed at the online meeting, and panellists will be asked to recommend outcomes to be used in the trial.

The conclusions of the expert panel will be shared with the patient and carer panel (below).

Patient and carer panel A patient and carer panel of people with a recent hospitalisation (<6 months) for HF will provide recommendations on trial endpoints. The patient-and-carer advisory group (PCAG) - a separate group - will also input into these discussions. This will ensure people with HF and their carers have a voice in the MAMS study design

Participants We will identify ~8-10 people to ensure we can achieve diversity of experience. Recruitment will be via current collaborators (BSH) and clinical co-applicants. People with a recent hospitalisation (<6 months) for severe congestion, or who have been an informal carer for such a person will be included.

Potential participants will be identified by each organisation and permission sought for their details to be passed to the researcher. Interested patients will be approached using both written invitations and discussions and written informed consent sought. Our PCAG members will also be able to join the group as participants if they wish.

Each eligible participant will be informed of the aims, methods, anticipated benefits and potential hazards of the study and their right to withdraw consent at any stage, using both the patient information sheet (PIS) and verbally. Patients will have the opportunity to ask any and all questions before giving written consent. Confirmation of the approach for study participation, outcome (participation or not) and confirmation of written consent will be documented in the medical notes by the study doctor.

Meeting content Three 90 minute online meetings will be used. Breaks will be built into meetings, and shorter meetings will be used if needed. Plain English summaries of the expert panel conclusions will be developed in collaboration with our person with HF co-applicant (LHD) and PCAG members to ensure materials are accessible.

Participants will be asked to share their thoughts on the adjunct treatments recommended by the expert panel e.g. concerns about identified side effects. A nominal group approach will be used to ensure all participants can contribute.60 Notes will be made of the discussions and decisions made and these will be shared after each meeting.

The final meeting (meeting 3) will focus on which outcome measures are important to the panel. The existing core outcome set and any additional outcomes identified by expert panel will be shared with the group, to ensure a range of outcomes are included for discussion. Participants will be invited to discuss all the possible outcomes and asked to rank their preferred outcomes.

Output Findings will be fed back to the research team. The PCAG and research team will decide upon the primary outcome based on the results of the expert panel and patient and carer panel work. Once the primary outcome has been chosen the expert panel will be reconvened by email to agree upon the minimal clinically important difference (MCID) and time-points at which to measure the primary outcome.

Once the number of interventions, the definition of usual care, the duration of treatment, the primary and secondary outcomes, and the minimal clinically important difference have been defined, the PCAG and research team will develop broad inclusion and exclusion criteria for the main trial which, in combination with the results of the online survey, will inform the statistical modelling (WP 2b).

ELIGIBILITY:
Inclusion Criteria:

1. Recent hospitalisation with heart failure (<6 months) or carer for a person with a recent hospitalisation with heart failure.
2. Able to participate in online group discussions in English

Exclusion Criteria:

1. Unable to participate in online group discussions in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See inclusion / exclusions
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Thematic Analysis of Nominal Group Discussions on Appropriate Endpoints for a Proposed Clinical Trial | From enrollment to end of third online monthly meeting (enrollment to 3 months)
  This qualitative study will use a nominal group technique to gather input from key stakeholders-including clinicians, researchers, and patient representatives-on appropriate endpoints for a proposed clinical trial. Participants will engage in structured group discussions guided by a topic guide with open-ended questions designed to prompt reflection on what makes an outcome meaningful, measurable, and feasible. Discussions will be audio-recorded, transcribed verbatim, and analyzed using thematic analysis. This process will involve inductive coding of the transcripts to identify recurring themes related to clinical relevance, patient-centeredness, feasibility, and scientific validity.
  After the discussions, participants will individually rank their preferred endpoints, supporting a structured consensus-building process. The combination of qualitative insights and ranked preferences will help prioritize outcomes that are both methodologically sound and aligned with stakeholder values.
Thematic Analysis of Nominal Group Discussions on which adjunctive therapies, at what dose, and for how long | From enrollment to end of third online monthly meeting (Enrolment to month 3)
  This qualitative outcome measure will be based on structured discussions using the nominal group technique to identify stakeholder perspectives on which adjunctive therapies should be used alongside the main intervention in a proposed clinical trial, including appropriate types, doses, and treatment durations. Participants-including clinicians, researchers, and patient representatives-will take part in guided sessions using a topic guide with open-ended questions. The discussions will be audio-recorded, transcribed verbatim, and analyzed using thematic analysis, which involves coding the data to identify key patterns and shared views.
  Themes will be developed around what therapies are considered beneficial, how dosing decisions should be made (e.g., based on weight, age, or clinical response), and what duration balances effectiveness with safety and feasibility. Participants will also rank their preferences after the discussion, enabling a consensus-driven prioritization of adjunctiv

CONTACTS AND LOCATIONS:
Overall Officials: Joe Cuthbert, MBBS MD, Principal Investigator — Wolfson Palliative Care Research Centre, Hull York Medical School, University of Hull, Cottingham Road, Kingston-Upon-Hull, HU6 7RX
Locations (1):
- Cardiology, Hull, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No